CLINICAL TRIAL: NCT07070921
Title: Assessing the Safety and Performance of the Novel CytaCoat Foley Catheter: A Prospective Randomized Controlled Study
Brief Title: Assessing Safety and Performance of the Novel CytaCoat Foley Catheter
Acronym: CYTA-FOL-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CytaCoat AB (Industry)
Collaborators: Sterimed Surgicals (India) Pvt Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CTRI/2025/05/086528
Record Dates: First submitted 2025-06-03; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Safety of the CytaCoat Foley Catheter; Performance of the CytaCoat Foley Catheter
Keywords: Safety; Performance; Biofilm; Adverse event; Fouling

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 to CytaCoat Foley catheter / Sterimed uncoated Foley catheter (15 subjects in each arm)
Who Masked: Outcomes Assessor
Masking Description: The healthcare practitioner placing the catheter will know the allocation (whether it is a CytaCoat Foley catheter or the comparator) but the subject will not know which catheter they have received. The healthcare practitioner removing the catheter may or may not know the allocation. Analyzed catheters for fouling / biofilm assessment will not state which arm the subject is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CytaCoat Foley catheter (Experimental): CytaCoat Foley catheters will be randomized 1:1 (15 patients in each arm), to patients in need of catheterization for 3 to 14 days.
  Interventions: Device: Foley catheter
- Sterimed uncoated Foley catheter (Active Comparator): Sterimed uncoated Foley catheters will be randomized 1:1 (15 patients in each arm), to patients in need of catheterization for 3 to 14 days.
  Interventions: Device: Foley catheter

INTERVENTIONS:
Device: Foley catheter — Drainage of urine from the bladder by transurethral catheterization with an indwelling Foley catheter of patients in need of a Foley catheter for 3 to 14 days.

SUMMARY:
This study is a prospective, single-center, single-blind, randomized, parallel assignment, controlled study to evaluate the safety and performance of the novel CytaCoat Foley catheter when compared to a Sterimed uncoated Foley catheter. Participants will include male and female adult subjects who require an indwelling urinary catheter for an expected duration of minimum 72 hours to 14 days.

The primary purpose of the clinical investigation is to determine whether the novel CytaCoat Foley catheter is safe to use in subjects. Safety is assessed by evaluation of adverse events (according to ISO 14155:2020).

The secondary objective is to assess the overall performance of the CytaCoat Foley catheter by evaluating usability experience by the healthcare personnel and subjects measured by using NRS (Numeric Rating Scale) scale.

Furthermore, the exploratory objective of this study is to assess for the presence of bacteriuria in urine and fouling / biofilm analysis of the used catheters.

DETAILED DESCRIPTION:
Study description This clinical study is designed to evaluate the safety and performance of the CytaCoat Foley catheter in subjects requiring urinary catheterization. The study will be conducted as a randomized, controlled trial with two parallel groups, wherein one group will receive the CytaCoat Foley catheter, and the other will receive a standard silicone Foley catheter as the control.

The study aims to determine the incidence of adverse events and to assess the overall performance of the CytaCoat Foley catheter in terms of patient outcomes, ease of use, and durability. The study will include patients who meet the inclusion criteria, with a defined follow-up period to assess the outcomes.

The primary purpose of the clinical study is to determine whether the novel CytaCoat Foley catheter is safe to use in subjects. The claims regarding clinical performance and clinical safety that the manufacturer intends to use:

* More comfortable
* Easy insertion and removal

Primary Objective The primary objective of this study is to determine the safety for the CytaCoat Foley catheter. Safety is assessed by evaluation of adverse events (according to ISO 14155:2020). Adverse events (AEs) and Serious Adverse Events (SAEs) are further divided into Adverse Device Effects (ADEs) and Serious ADEs (SADEs).

Secondary Objective The secondary objective is to assess the overall performance of the CytaCoat Foley catheter by evaluating usability experience by the healthcare personnel and subjects measured by using NRS scale.

1. Assessment of usability of the Foley catheter by a responsible nurse/physician with the NRS scale (0-10) using a questionnaire.
2. Assessment immediately after removal of the catheter of pain, irritation, and discomfort measured with the NRS scale (0-10) using a questionnaire asking subjects about their experience using the catheter.
3. Telephonic follow-up assessment between 7±1 days after removal of the catheter using a questionnaire asking subjects about their experience using the catheter.

Furthermore, the exploratory objective of this study is to assess for the presence of bacteria in urine and fouling / biofilm analysis of the used catheter.

This study is a prospective, single-center, single-blind, randomized, parallel assignment, controlled study to evaluate the safety and performance of the novel CytaCoat Foley catheter when compared to a Sterimed uncoated Foley catheter.

The estimated enrolment is 30 subjects, randomized 1:1 to CytaCoat Foley catheter / Sterimed uncoated Foley catheter (15 subjects in each arm).

In this study, the duration of catheterization is a minimum of 72 hours and a maximum of 14 days. During this period assessments of each subject shall be recorded in the CRF on the day of catheterization (day 0) and day of catheter removal. There is a telephonic follow-up between 7±1 days after the removal of the catheter, which shall be recorded in the CRF (Case Report Form). The data of the urine analysis / culture report and the fouling / biofilm data shall be updated in the CRF after receiving it.

Description of clinical study-related procedures Each subject will take part in the clinical study from the time the subject/legal representative signs the ICF (Informed Consent Form).

APACHE II score is a general measure of disease severity based on current physiological measurements, age & previous health conditions. The score can help in the assessment of subjects to determine the level & degree of diagnostic & therapeutic intervention. APACHE II score (Acute Physiology And Chronic Health Evaluation) will be used to compare baseline characteristics in subjects recruited from critical care. Critically ill subjects will be excluded from this clinical study based on the result obtained from the APACHE II score assessment. Subjects having APACHE II scores more than or equal to 28 will not be considered for the clinical study.

Subjects will be screened using a urine dip stick for presence of bacteriuria. A urine culture will be sent if found positive for bacteriuria. The presence of one or more species of bacteria growing in the urine at specified quantitative counts (≥10^5 Colony Forming Units [CFU]/mL) will be defined as bacteriuria in urine culture.

After the screening, the subjects will be block randomized to either a CytaCoat Foley catheter or a Sterimed uncoated Foley catheter. Subjects will be assigned to receive trial treatment, catheterization for at least 72 hours and up to 14 days or until the catheter has been removed as per standard hospital guidelines, the investigator's decision to withdraw the subject, noncompliance with trial treatment or procedures, unacceptable adverse event, or the subject withdraws consent.

Healthcare providers and the subjects will be asked to complete questionnaires provided in the CRF.

Prior to removing the urinary catheter, a urine culture will be sent for analysis. For this purpose, the catheter between the patient and the drainage bag will be clamped for 30 minutes to allow fresh urine to accumulate in the bladder. During this period, the sampling port on the catheter will be identified and sterilized using an antiseptic wipe, allowing it to air dry completely. After the 30-minute interval, a sterile syringe will be attached to the sampling port, and a volume of 10-20 mL of urine will be carefully aspirated. The collected urine will then be transferred into a labelled sterile culture container.

All indwelling catheters will be sent for fouling / biofilm examination after the removal, according to a provided method description (50).

A subject data sheet will be used to collect subject demographic data, a questionnaire will be used to capture the safety, comfort, and complications related to the catheter.

A telephonic follow-up will be performed by the study nurse 7±1 days after removing the study catheter.

Monitoring The clinical study will be monitored by an independent monitor before the clinical study begins, during the clinical study, and after the clinical study has been completed, so as to ensure that the clinical study is carried out according to the clinical study protocol and that data is collected, documented, and reported according to ISO 14155:2020 and applicable ethical and regulatory requirements. Monitoring is intended to ensure that the subject's rights, safety, and well-being are met as well as data in the CRF are complete, correct, and consistent with the source data.

Study devices The uncoated Sterimed catheter is made from 100% medical grade silicone and is suitable for subjects requiring in-dwelling catheterization.

The CytaCoat Catheter is made of a silicone Foley balloon 2-way catheter from Sterimed, coated with a CytaCoat coating applied to both the inside and the outside of the catheter and the balloon. The coating of the device reduces the friction of the catheter surface to the bladder and urethra, enhancing subject comfort on insertion, carriership and withdrawal.

The coating reduces fouling, prevents biofilm (EPS, Extracellular Polymeric Substances) formation and subsequent encrustation. The mode of action of the coating is based on a super hydrophilic surface and a covalently bonded anti-fouling ligand. This prevents the build-up of dead bacteria on the device surface and retains its effectiveness throughout extended use.

The coating does not elute toxins or an active antimicrobial agent. The healthy microbial flora is therefore not disturbed by the use of the catheter.

The intended clinical benefits and performance:

1. Drainage of urine from the bladder.
2. Ability to stay in place and offer consistent drainage.
3. Flexible tube which can easily pass through the urethra.
4. Comfort on insertion, carriership, and withdrawal of the catheter.
5. Helpful for monitoring the urine output of the subject.
6. Reduction of fouling and biofilm formation during catheterization and carriership.

Final outcome parameters (for commercial product):

* Ease of use.
* Comfortable during usage, cause less pain and discomfort.
* Less incidence of fouling and biofilm formation.

Claims regarding clinical performance and clinical safety that the manufacturer intends to use:

* Less discomfort.
* Easy insertion and removal for the subject.
* Easy insertion and removal for the healthcare provider.

ELIGIBILITY:
Inclusion Criteria:

* Adults, male and female, aged 18 to 84 years
* Subjects in need of a urinary catheter for a minimum of 72 hours
* Subjects who can accommodate a size of 14, 16 and 18 French Foley catheter
* Written informed consent
* Subject to be conscious

Exclusion Criteria:

* Pregnant or breastfeeding women
* Critically ill subjects with a life-threatening disorder (Subjects having an APACHE II score ≥ 28)
* Subject with a known silicone allergy or sensitivity
* Previous enrolment in the present study
* Simultaneous participation in another clinical study that may impact the primary endpoint
* Subject with pre-existing urinary catheter for more than 48 hours
* Subject with symptomatic genitourinary pathology
* Expected severe non-compliance to the protocol as judged by the principal investigator

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of Safety through incidence of adverse events and serious adverse events of the CytaCoat Foley catheter. | 3 - 14 days
  Adverse events (AEs) and serious adverse events (SAEs) which are further divided into adverse device effects (ADEs) and serious ADEs (SADEs) will be assessed.

SECONDARY OUTCOMES:
Assessment of the overall performance related to the CytaCoat Foley catheter using questionnaires. | 3 - 14 days
  Assessment of the overall performance related to the medical device based on Foley catheter usability experience by the healthcare personnel and subjects will be performed using questionnaires with the NRS scale (0-10) by the responsible nurse/physician, and by the subjects immediately after removal of the catheter and after 7±1 days after removal.

OTHER OUTCOMES:
Microbiological assessment of the catheter after use | 3 - 14 days
  To assess for the presence of bacteriuria in urine and fouling / biofilm analysis of the used catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Soumya Madhusudhan, MD, Principal Investigator — Department of Neuro ICU, St John's Medical College Hospital
Locations (1):
- St. John's Medical College Hospital, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No